CLINICAL TRIAL: NCT02663310
Title: Surgical Decompression/Untethering Combined With Weight Bearing Rehabilitation in Chronic Spinal Cord Injury Subjects
Brief Title: Treatment for Chronic Spinal Cord Injury: Surgery With Rehabilitation vs Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kunming Tongren Hospital (Industry)
Collaborators: Hong Kong Spinal Cord Injury Fund (Unknown); China Spinal Cord Injury Network (Network)
Responsible Party: Principal Investigator, Hui Zhu, Director, Kunming Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KunmingTH_HZ_001
Record Dates: First submitted 2015-12-28; First posted 2016-01-26 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; Kunming Locomotor Scale; surgical decompression; untethering; weight bearing rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Surgical Procedures, Operative; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery with Rehabilitation (Experimental): Surgically removed cysts, and collected intracystic fluids and cerebrospinal fluid for histological and molecular analyses. Samples will be collected during the surgery and will be cryo-protected for further analyses. All subjects will enroll for intensive rehabilitation 60 days after surgery.
  Interventions: Procedure: Surgery; Procedure: Rehabilitation
- Rehabilitation (Active Comparator): All subjects will enroll for intensive rehabilitation everyday as instruction.
  Interventions: Procedure: Rehabilitation

INTERVENTIONS:
Procedure: Surgery — Surgery treatment of the injured vertebra(e), internal fixation of the vertebral column, and bilateral laminectomy for epidural decompression were followed directly by neurosurgical management, including separation of the arachnoid adhesion to restore cerebrospinal fluid flow and debridement of the spinal cord necrotic tissue with concomitant intramedullary decompression.
  Arms: Surgery with Rehabilitation
Procedure: Rehabilitation — The patients need to do intensive rehabilitation everyday. （1）The limb comprehensive training is Kunming Locomotor exercise, 60 minutes twice per day.(2)The exercise therapy includes sit-ups by 30 times, twice per day; half bridge exercise by 10 times, twice per day; backward flight movement by 10 times, twice per day; sling exercise training by 30 minutes, twice per day; and postural transfer functional training by 10 minutes, twice per day. (3)The balance training include ball toss training by 10 minutes, twice per day; and balance board training by 10 minutes, twice per day. (4)The wheelchair training will be taken 20 minutes each, twice per day. (5)The isokinetic training needs to perform 20 minutes each, twice per day.

SUMMARY:
The purpose of this study is to investigate the efficacy of surgical decompression/untethering, combined with weight bearing rehabilitation, on neurological recovery following chronic spinal cord injury.

DETAILED DESCRIPTION:
Safety Issues:

Safety issues need to be watched are: occurrence of known and unknown undesirable incidences, moving up injury levels, loss of previously preserved neurological functions, vital physical signs, and worsening of EKG and lab results. If unforeseen issues occur, patients will be consulted to determine whether treatments will be continued.

Adverse events:

Adverse events may occur during the trail and these events will be recorded. The severity of the events and their relationship to the experimental therapy will be determined, documented and reported to the Data Monitoring and Safety Committee who will determine how these events will be handled if they occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult subjects, 18-60 years of age
* Have a clinical diagnosis of chronic spinal cord injury (≥ 12 months after traumatic spinal cord injury).
* Neurological examination: ASIA-A
* Injury levels: T1-T12 spinal levels
* The diagnosis of spinal cord injury is confirmed by MRI
* Subjects must be able to read, write and complete visual analogue scale
* Voluntarily signs and dates an informed Consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures. If a subject consents to participation but is not in a position to personally sign and date the informed consent form because of his or her physical condition, the consent must be confirmed at the time of consent orally, signed on behalf by the subject's relative, and by an impartial witness who is present throughout the whole informed consent process.

Exclusion Criteria:

* Severe head injury
* Subjects with severe osteoporosis or joint diseases
* Subjects with severe pressure sore
* Sign of kidney, cardiovascular, liver disorders
* Subjects with internal medical and/or infectious diseases (including but not limited to Hepatitis B and HIV carriers)
* Pregnant women or women at lactation stages
* Medically or mentally unstable according to the judgment of the investigator
* History of multiple sclerosis or peripheral demyelination
* Any criteria which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change of Kunming Locomotor Scale in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  Kunming Locomotor Scale is a 10-grade Roman numeral locomotion scoring system. Grade I, the patient can not stand; grade II, the patient was able to stand with weight support and help in fixing the knee; grade III, the patient was able to stand with weight support; grade IV, the patient was able to walk with wheeled weight support and help in fixing the knee of the weight bearing leg; grade V, the patient was able to walk with wheeled weight support; grade VI, the patient was able to walk with the help of a light four-leg support; grade VII, the patient was able to walk with a pair of crutches; grade VIII, the patient was able to walk with a cane; grade IX, the patient was able to walk without support but staggeringly; and grade X, the patient was able to walk stably without support.

SECONDARY OUTCOMES:
Change of Walking Index for Spinal Cord Injury in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  The Walking Index for Spinal Cord Injury evaluates the amount of physical assistance, braces or devices required to walk at 10 meters.
Change of Spinal Cord Independence Measure in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  The Spinal Cord Independence Measure assesses patients' self-care, respiration and sphincter management, and mobility abilities with a total score of zero to 100.
Change of American Spinal Injury Association Impairment Scale in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  American Spinal Injury Association Impairment Scale as international standards for neurological classification of spinal cord injury, is a 5 point ordinal scale to identify patient's sensory and motor levels, from A (complete SCI) to E (normal sensory and motor function).
Change of Modified Ashworth Scale in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  Modified Ashworth Scale is considered the primary clinical measure of muscle spasticity in patients with neurological conditions, with Grade of 0, 1, 1+, 2, 3 and 4 (from no increase in muscle tone to affected parts rigid in flexion or extension).
Change of Numerical Rating Scale in 1 year | Day 0, Day 15, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and 1 year
  The Numerical Rating Scale is to assess pain intensity in patients who are able to self report ranging from 0 (no pain) to 10(unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhu, MD, Principal Investigator — Kunming Tongren Hospital
Locations (1):
- Kunming Tongren Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu H, Guest JD, Dunlop S, Xie JX, Gao S, Luo Z, Springer JE, Wu W, Young W, Poon WS, Liu S, Gao H, Yu T, Wang D, Zhou L, Wu S, Zhong L, Niu F, Wang X, Liu Y, So KF, Xu XM. Surgical intervention combined with weight-bearing walking training promotes recovery in patients with chronic spinal cord injury: a randomized controlled study. Neural Regen Res. 2024 Dec 1;19(12):2773-2784. doi: 10.4103/NRR.NRR-D-23-01198. Epub 2024 Jan 31. PMID 38595294
- See also: International Spinal Cord Injury Treatment Center, Kunming Tongren Hospital — http://en.kmtrh.org/